CLINICAL TRIAL: NCT02390648
Title: Efficacy of Ginger as an Adjunctive Prophylaxis for Chemotherapy-induced Nausea and Vomiting: Randomised Double-blind Placebo-control Cross Over Study
Brief Title: Efficacy of Ginger as an Adjunctive Prophylaxis for Chemotherapy-induced Nausea and Vomiting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 732/2557(EC1)
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — ginger extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ginger (Experimental): Ginger capsule (500 mg) taking twice a day by mouth during the first 5 days of chemotherapy cycle
  Interventions: Drug: Ginger
- Placebo (Placebo Comparator): Placebo capsule taking twice a day by mouth during the first 5 days of chemotherapy cycle
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ginger — Ginger capsule (500 mg) taking twice a day by mouth during the first 5 days of chemotherapy cycle
  Arms: Ginger
Drug: Placebo — Placebo capsule taking twice a day by mouth during the first 5 days of chemotherapy cycle
  Arms: Placebo

SUMMARY:
Breast cancer patient receiving AC regimen chemotherapy (Doxorubicin + Cyclophosphamide) who has nausea score from 40/100 VAS or vomiting after the first or second cycle of chemotherapy is recruited. The patient who meets the eligibility criteria and provides informed consent is randomised to receive either Ginger capsule (500 mg) or placebo taking twice a day by mouth during the first 5 days of chemotherapy cycle. The study drug will be switched on the subsequent cycle (i.e. the patient who received Ginger capsule will receive placebo and vice versa). The primary outcome is the nausea score and vomiting during the first 5 days of each chemotherapy cycle when receiving the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed breast cancer patient
* Received AC regimen chemotherapy (Doxorubicin + Cyclophosphamide) and has nausea score at least 40/100 VAS or has vomiting
* Expect to receive at least 2 further cycles of AC regimen chemotherapy
* Provide informed consent

Exclusion Criteria:

* Pregnancy or lactation
* Has nausea or vomiting during 24 hours before chemotherapy
* Has other causes of nausea or vomiting eg. brain metastasis, gut obstruction, hepatitis or recent abdominal or pelvic irradiation within 1 week before chemotherapy
* Received any chemotherapy regimen other than AC regimen
* Allergic or intolerance to ginger

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Nausea score | The first 5 days of chemotherapy cycle

CONTACTS AND LOCATIONS:
Overall Officials: Nopadol Soparattanapaisarn, MD, Principal Investigator — Lecturer
Locations (1):
- Siriraj Hospital, Bangkok, Thailand